CLINICAL TRIAL: NCT02398162
Title: The Natural Immune Response In Pediatric Scrub Typhus In Chiangrai
Brief Title: Scrub Typhus Pediatric Immunology Study
Acronym: NIRPS
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Li Ka Shing Foundation (Other); Mahidol University (Other); Chiangrai Prachanukroh Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MICRO1402
Record Dates: First submitted 2015-02-27; First posted 2015-03-25 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Scrub Typhus
Keywords: Scrub Typhus in Pediatric; Immunology
MeSH Terms: conditions — Scrub Typhus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- STP: Scrub Typhus Patients (STP, n=60) Cohort. Blood samples will be collected at baseline (the day of presentation to hospital), 2 weeks later in hospital, 12 weeks after baseline at the clinic visit and 1 year later. Data on clinical presentation and relapses will be recorded. Eschar swab specimens and a non-invasive specimen of the dark crust will be also collected from STP group on the day of enrollment.
  Interventions: Procedure: Multi Blood Collections
- STE: Scrub Typhus Exposed (STE, n=80) Cohort. Single blood sample collection.
  Interventions: Procedure: Single Blood Collection
- STH: Scrub Typhus Healthy (STH, n=30) Cohort. Single blood sample collection
  Interventions: Procedure: Single Blood Collection

INTERVENTIONS:
Procedure: Multi Blood Collections — At baseline (the day of presentation to hospital), 2 weeks, 12 weeks and 1 year later.
  Groups: STP
Procedure: Single Blood Collection — On the enrollment day
  Groups: STE; STH

SUMMARY:
This is an observational study of the natural immune response to scrub typhus in patients recruited from Chiangrai Prachanukroh Hospital, N-Thailand. Febrile patients with a positive IgM rapid diagnostic test will be asked if they wish to take part in a study to improve the understanding of how the body responds to scrub typhus. Blood samples will be collected from each participant ("STP", n=60) at baseline (the day of presentation to hospital), 2 weeks later in hospital, 12 weeks after baseline at the clinic visit and 1 year later. Data on clinical presentation and relapses will be recorded. Control subjects are scrub typhus exposed patients from a rural village in the caption area of Prachanukroh Hospital ("STE", n=80; approx. 40 children and 40 adults), and healthy adults blood donors from Bangkok ("STH" n=30) - these subjects will be enrolled for one single blood sample. The study team will also collect eschar swab specimens from STP group and a non-invasive specimen of the dark crust on the day of enrollment.

Funder: Li Ka Shing Foundation [Grant C13004]

DETAILED DESCRIPTION:
Primary Objective:

o To measure and characterize the memory and effector T-cell responses, as well as the humoral response in young patients with acute scrub typhus and to compare theseThese acute responses will be compared to responses in the convalescent phase of the same individuals at 2, 12 and 52 weeks later, as well as to scrub typhus-exposed controls and to healthy controls.

Secondary Objectives:

* To establish ELISpot and flow cytometer based immunology assays using human samples collected in rural areas of high scrub typhus endemicity.
* To set up a prospective cohort study of paediatric scrub typhus in a region of high endemicity

Description of the Study Sites and Population Chiangrai Prachanukroh Hospital in Chiangrai province, N-Thailand is ideally suited for this study. We have a well-established collaboration, due to a previously completed multi-year fever study and an excellent relationship with local senior doctors, staff and the hospital-based laboratory. There is a very high rate of scrub typhus cases admitted to the infectious diseases ward and the recent establishment of a MORU (Mahidol Oxford Tropical Medicine Research Unit) satellite laboratory within the hospital facilities, make this study site unique and highly suited for performing this research project. This study will contribute significantly towards the long-term aim of developing the Chiangrai study site towards an immunogenicity monitoring field site for vaccine trials.

The 'scrub typhus' patients (STP) are febrile children recruited from the ID and/or pediatric wards at Prachanukroh hospital during an acute hospitalization due to scrub typhus, and followed up as described above.

The scrub typhus 'exposed' cohort (STE) will consist of children and adults recruited from two villages in an area where scrub typhus is reported as a common disease. This cohort has a high risk of previous contact with scrub typhus, and it is unknown if they had an asymptomatic or sub-clinical infection in the past, but we expect the presence of some form of immune memory regarding cellular and/or humoral immunity in a large proportion of these subjects.

The healthy scrub typhus naïve control group (STH) does not necessarily need to include children, as the principle is to compare a non-exposed immune response to previously exposed and/or acute cellular responses. Thus, the 'Healthy Cohort' will be recruited from the staff at MORU and/or the Faculty of Tropical Medicine in Bangkok.

ELIGIBILITY:
Inclusion Criteria:

Scrub Typhus Patients (STP) Cohort inclusion criteria

* Age >6 months to ≤18 years (STP consist of pediatrics only)
* Scrub Typhus Rapid test positivity (SDm Standard Diagnostics RDT, Korea)
* O. tsutsugamushi PCR-positivity (if PCR capability is available by the start of the study)
* Fever in ≤ 14 days of presentation to Hospital
* Willingness to participate in the study and written informed assent previously obtained from the patient, and written informed consent obtained from the patient's parent(s), guardian(s) or representative(s)

Scrub Typhus Exposed (STE) Cohort inclusion criteria

* Age >6 months to ≤18 years and age >18 years (STE consist of paediatrics and adult )
* Historical diagnosis of scrub typhus, as defined by rapid diagnostic test, serology and/or PCR positivity (more than 2 years ago), or living in an endemic area with high risk of previous exposure.
* Currently well and healthy
* Willingness to participate in the study and written informed assent previously obtained from the patient, and written informed consent obtained from the patient's parent(s), guardian(s) or representative(s)

Scrub Typhus Healthy (STH) Cohorts inclusion criteria

* Age >18 years (STH consist of adults only)
* Currently well, no medical problems requiring hospital specialist supervision
* Willingness to participate in the study and written, informed consent previously obtained
* Residing in Bangkok for at least the 2 past recent years

Exclusion Criteria:

Scrub Typhus Patients (STP) Cohort exclusion criteria:

* Current TB or TB treatment in ≤ 6 months (contains Orientia-effective antimicrobial)
* Documented HIV infection, use of steroids, chemotherapy, other immunosuppressant therapy or herbal remedies containing steroids and/or pregnancy

Scrub Typhus Exposed (STE) Cohort exclusion criteria:

* Significant acute intercurrent illness at the time of blood draw including fever >37.5°C or infection (including TB) requiring antibiotics
* Documented HIV infection, use of steroids, chemotherapy, other immunosuppressant therapy or herbal remedies containing steroids and/or pregnancy

Scrub Typhus Healthy (STH) Cohorts exclusion criteria:

* Previous history of scrub typhus
* Significant acute intercurrent illness at the time of blood draw including fever >37.5°C or infection (including TB) requiring antibiotics
* Documented HIV infection, use of steroids, chemotherapy, other immunosuppressant therapy or herbal remedies containing steroids and/or pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Cases: Male and female patients ≤ 18 years of age with acute scrub typhus (n=60). Controls: people exposed to scrub typhus (approx. 40 children and 40 adults from Chiangrai, total n=80) preferably age-matched, healthy and non-febrile, and healthy adult scrub typhus-naïve controls from Bangkok (n=30), total n=170.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Cellular immune response to Orientia tsutsugamushi | 2 years
  Characterize the cellular immune response to Orientia tsutsugamushi, based on immune cell phenotyping and quantitation of effector, memory & regulatory T cell functions.

SECONDARY OUTCOMES:
T-cell subsets during the scrub typhus infection | 2 years
  Identification of T-cell subsets affected by apoptosis during the course of acute scrub typhus.
Antibody isotypes during the scrub typhus infection | 2 years
  Determination of the antibody isotypes and their dynamics involved in natural scrub typhus infection.
Adaptive immune response to Orientia tsutsugamushi | 2 years
  Characterisation of the adaptive immune response to Orientia tsutsugamushi, measured by ex vivo interferon-gamma ELISPOT in spot forming cells per million peripheral blood mononuclear cells (SFC/106PBMC), using four Orientia antigens (whole cell antigen, 56kDa, 47kDa and scaC) in samples of acute disease and long term follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Daniel Paris, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (1):
- Chiangrai Prachanukroh Hospital, Chiang Rai, Thailand